CLINICAL TRIAL: NCT03039231
Title: Investigation of the Freespira Breathing System in the Treatment of PTSD
Brief Title: Investigation of the Freespira Breathing System in the Treatment of Post Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Health Sciences, Inc. (Industry)
Collaborators: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-16-FS02
Record Dates: First submitted 2017-01-25; First posted 2017-02-01 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2018-04

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Freespira Breathing System (FBS) (Experimental): The Freespira Breathing System (FBS) developed by Palo Alto Health Sciences, Inc, is a portable home device used for breathing biofeedback in adults with panic disorder (PD). FBS has received FDA clearance for the treatment of PD adults and is currently commercially available with more than 150 therapist providing the treatment nationally. FBS has not yet been tested for efficacy in an adult post traumatic stress disorder (PTSD) population. It has been suggested that there is overlap in the presence and persistence of symptoms between PD and PTSD patients. The primary goal of this study is to determine whether the FBS will produce similar benefit (both in quality and magnitude) in the defined population of patients with PTSD.
  Interventions: Device: Freespira Breathing System

INTERVENTIONS:
Device: Freespira Breathing System — Following authorization from a study team member, patient will be assigned an FBS to take home and perform 4 weeks of training exercises twice a day for 17 minutes each time. Efficacy of the FBS system will be evaluate over the 4 week period and at 2 and 6 month follow-up periods.

SUMMARY:
This study will test the efficacy of the Freespira Breathing System in adults with post traumatic stress disorder (PTSD).

DETAILED DESCRIPTION:
The Freespira Breathing System (FBS) developed by Palo Alto Health Sciences, Inc, is a portable home device , and has been employed in breathing biofeedback in adults with panic disorder (PD). The FBS has received FDA clearance for the treatment of PD adults and is currently commercially available.

This study is a prospective, single arm, un-blinded investigation of the Freespira Breathing System in the PTSD population.

ELIGIBILITY:
Inclusion Criteria:

Note: Office visits required. Patients must live locally in San Francisco/Silicon Valley Bay Area to participate.

Patients with a primary diagnosis of PTSD

* Additional DSM-V disorders are acceptable and will be documented.

  * Subjects over 18 years of age
  * Subjects with a Clinician's Global Impression (CGI-S) score of ≥ 4
  * Subjects with a CAPS-5 score of ≥ 30
  * If on psychotropic medication(s), on a stable dose during the course of treatment
* This can include benzodiazepine use that is prescribed on an as needed basis. • If on psychotropic medication(s), patient agreement to maintain their current stable dose from point of study entry until the 2-month post-treatment assessment.

Exclusion Criteria:

* Subject is pregnant.
* Current enrollment in another device or drug study.
* Enrollment in another drug or device study that is not at least 30 days past the final follow-up visit.
* Currently undergoing cognitive behavioral therapy, or equivalent that is focused addressing PTSD including any evidenced based therapy that focuses on PTSD, including cognitive processing therapy, EMDR, prolonged exposure therapy, Virtual reality therapy, during trial and 2 month follow up. Cognitive therapy must be discontinued 1 month prior to enrolling in this study.
* Severe suicidality, in the judgment of the interviewer and taking the CHART assessment into account
* Psychotic disorder diagnosis, including schizophrenia and schizoaffective disorder
* Presence of uncontrolled bipolar disorder as described below -

  * The subject has experienced a manic episode in the past 6 months and is not considered under control by reviewer
  * Bipolar disorder is considered the primary diagnosis for the subject, in the interviewer's opinion.
* No Alcohol, drug use disorder that requires medical treatment . If stable under medical supervision treatment for drug/alcohol use, then OK
* Cardiovascular or pulmonary disease, such as COPD.

  * Score of ≥ 10 on the COPD assessment
  * EtCO2 of ≥ 48 mmHg at first treatment visit
* Epilepsy or seizures
* Inability to understand or comply with study procedures.
* The investigator feels that for any reason the subject is not eligible to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-08-25 (Actual)

PRIMARY OUTCOMES:
Primary outcome of this study will be quantitative improvements using the Clinician Administered PTSD Scale (CAPS - 5). | 2 month and 6 months post treatment
  Using this scale, Response is defined as a reduction of 6 or more points. Remission is defined as Response plus no longer meeting clinical symptom criteria and having a severity score < 25.

SECONDARY OUTCOMES:
Change in Patient Health Questionnaire (PHQ-9) Score | 2 month and 6 months post treatment
  Change in condition (score) as recorded from baseline
Change in 36-Item Short Form Survey (SF-36) Score | 2 month and 6 months post treatment
  Change in condition (score) as recorded from baseline
Change in Clinical Global Impression (CGC-S) Score | 2 month and 6 months post treatment
  Change in condition (score) as recorded from baseline
Change in Panic Disorder and Severity Scale (PDSS) Score | 2 month and 6 months post treatment
  Proportion achieving a clinically significant 40% decrease, proportion achieving a remission score <= 5.
Proportion achieving "Remission" by CAPS-5 Score | 2 month and 6 months post treatment
  Remission is defined as 'Response' plus no longer meeting clinical symptom criteria and having a severity score of <25.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Ostacher, MD, Principal Investigator — VA Palo Alto Health Care System
Locations (1):
- Stanford University School of Medicine/Palo Alto Veterans Institute for Research, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ostacher MJ, Fischer E, Bowen ER, Lyu J, Robbins DJ, Suppes T. Investigation of a Capnometry Guided Respiratory Intervention in the Treatment of Posttraumatic Stress Disorder. Appl Psychophysiol Biofeedback. 2021 Dec;46(4):367-376. doi: 10.1007/s10484-021-09521-3. PMID 34468913
- See also: For more information about the Freespira Breathing System click on link — http://www.freespira.com